CLINICAL TRIAL: NCT05660499
Title: Assessment of the Presence of Symptoms of End-of-life Discomfort and Their Management in Children With a Primary Brain Tumor in the Grand Est Region. Impact of the Development of Pediatric Palliative Care
Brief Title: Impact of the Development of Pediatric Palliative Care
Acronym: PTB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8137
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Primary Brain Tumor
Keywords: Primary Brain Tumor; Pediatric Palliative Care
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite medical advances, cancer remains the leading cause of death by disease in children.

Brain tumors are the second most common cause of cancer in children after leukemia, representing 25% of pediatric cancers.

The overall survival rate is about 50% with extremes ranging from less than 5% to more than 90% depending on the histological type of brain tumor.

The end of life of children with a brain tumor is marked by the possibility of discomfort symptoms, painful or not, and by a progressive neurological deterioration, which makes the management of these children complex for both families and health professionals.

Over the last decade, the concept of palliative care has been increasingly integrated into pediatric onco-hematology services with the primary objective of better symptom control in a global approach to the child and his or her family in order to aim at a better quality of life.

DETAILED DESCRIPTION:
The main objective of the study is to compare the occurrence and management of end-of-life symptoms in children who died of a primary brain tumor over 2 periods, in 2009 - 2010 and in 2019 - 2020, followed in the Pediatric Oncology departments of Strasbourg, Besançon, Dijon, Nancy and Reims.

ELIGIBILITY:
Inclusion criteria:

* Patient less than 17 years of age
* Suffering from a primary brain tumor
* Died during the period 2009-2010 or during the period 2019-2020
* Follow-up in one of the Pediatric Oncology departments participating in the study (Strasbourg, Besançon, Dijon, Nancy and Reims)
* Absence of refusal expressed in the medical file by the parents or the holder(s) of parental authority concerning the reuse of the child's personal data for research purposes.

Exclusion criteria:

* Refusal expressed in the medical file by the parents or the holder(s) of parental authority concerning the reuse of the child's personal data for research purposes
* Patient with a brain tumor secondary to another cancer

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: - Patient less than 17 years of age suffering from a primary brain tumor
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence of symptoms of physical or psychological discomfort in the last 4 months of life | up to the last 4 months of life

CONTACTS AND LOCATIONS:
Locations (1):
- Service de soins Palliatifs - CHU de Strasbourg - France, Strasbourg, France